CLINICAL TRIAL: NCT07145671
Title: The COCCOS Study: Implementing and Evaluating a Transition Program for Young Persons With Chronic Conditions
Brief Title: The COCCOS Study: a Transition Program for Young Persons With Chronic Conditions
Acronym: COCCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Ghent (Other); University Hospital, Ghent (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Eva Goossens, professor, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B3002024000166; G066622N (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2025-06-26; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus; Obesity; Asthma
Keywords: adolescent; young adult; transitional care; transition program
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition program (Experimental): A transition program (TP) was developed, as part of the first work package of the COCCOS project, in close collaboration with stakeholders (i.e., AYA patients, parents and HCPs) based on participatory action research methods (i.e., Experience-Based Co Design, including photovoice). Based on this study, the developed TP entailed four key moments: (i) a transition consultation, (ii) a consultation without parents, (iii) a joint consultation, and (iv) a feedback moment. Over a course of approximately 9-15 months (this can differ considering different pathologies have different care trajectories (e.g., frequency of consultations)), AYAs will receive an intensive person-centered transition program consisting of the four key moments.
  Interventions: Other: Transition program
- Standard care (No Intervention): Participants in this arm will receive standard of care.

INTERVENTIONS:
Other: Transition program — Transition Consultation:
  Pediatric HCP introduces the transition process to AYA and family. A contact person is assigned (ideally the AYA's trusted HCP), along with someone from the AYA's personal network. Key points are recorded in the Individualized Transition Plan (ITP).
  Independent Visit:
  AYA has a solo consultation (parents briefly step out). They complete the Ready Steady Go checklist. The ITP is updated, and concerns are discussed.
  Joint Consultation:
  Pediatric and adult HCPs meet with the AYA. A new adult contact is assigned, and the AYA picks a pediatric contact for feedback. Checklist is completed again.
  Feedback Moment:
  After transfer, the pediatric contact checks in. The checklist guides discussion; feedback is shared across teams, and follow-up arranged if needed.
  Arms: Transition program

SUMMARY:
A study is undertaken to examine the feasibility of the newly developed transition program in adolescents with type 1 diabetes, asthma and obesity in a multicentric setting. Specific objectives for this study are: (1) examining the impact of the program in terms of patient-reported health outcomes, (2) examining patients' and healthcare providers' experiences related to the program implementation process, and (3) examining the impact of the program in terms of cost-effectiveness.

DETAILED DESCRIPTION:
Chronic conditions are increasingly common in youth, with 10-25% affected and over 85% reaching adulthood. This rise stems from higher incidence of conditions like diabetes and improved survival of congenital diseases. These young patients face a lifelong risk of complications, requiring continuous, age-appropriate care. A well-managed transfer from pediatric to adult care is essential, yet up to half of adolescents lack adequate preparation. Poor transitions can lead to care disruption, worse health outcomes, and higher costs. Structured transition programs (TPs) can improve self-management, adherence, and health outcomes, while reducing costs. However, implementation and long-term integration of TPs remain limited, especially for common chronic conditions. Following the development of a TP through Experience-Based Co-Design in the COCCOS project, the next phase involves a feasibility study to assess its preliminary impact.

A multicenter, quasi-experimental pre-test post-test study will assess a co-designed transition program at two Belgian hospitals (UZA and UZ Ghent), comparing it to usual care. AYAs aged 17-18 with type 1 diabetes, asthma, or obesity will be recruited (n=150). The intervention group will receive the TP over 9-15 months; the control group (CG) will receive usual care. Assessments occur at baseline, transfer, and 4 months post-transfer.

The TP includes four stages:

1. Transition consultation (intro to transition and planning)
2. Independent visit (AYAs attend without parents, guided by Ready Steady Go-checklist)
3. Joint consultation (with pediatric and adult HCPs)
4. Feedback moment (post-transfer evaluation) An individualized transition plan (ITP) will be created and used throughout the TP. This ITP will be available via hospital portals, where AYAs can review and update their plan as needed.

The primary outcome of the study is transition readiness, measured using the Transition Readiness Assessment Questionnaire (TRAQ). Secondary outcomes include patient empowerment (GYPES), medication adherence (MMAS), quality of life (EQ-5D-5L), and anxiety and depression (HADS). Clinical indicators such as emergency visits, missed consultations, and disease-specific biomarkers will also be collected. Data will be analyzed using descriptive statistics, paired and independent t-tests, and multivariable regression analyses. To account for baseline differences between groups, inverse probability treatment weighting (IPTW) will be applied. Significance will be set at p < 0.05. A process evaluation will be conducted alongside the effect evaluation to understand how the TP was implemented and received by AYAs, families, and healthcare providers. Data will be gathered using observations, satisfaction questionnaires, and semi-structured interviews. Evaluation will focus on fidelity, dose delivered and received, reach, contextual influences, and any adaptations made during the intervention. Qualitative data will be analyzed thematically using NVivo software. The cost-effectiveness of the TP will be assessed using a health economic model, developed in accordance with ISPOR guidelines. Cost data will include implementation expenses and healthcare utilization, while effectiveness data will focus on quality-adjusted life years (QALYs) derived from the EQ-5D-5L. The model will calculate an incremental cost-effectiveness ratio (ICER) comparing the TP with usual care. Sensitivity analyses and bootstrapping will be performed to address uncertainty, and cost-effectiveness acceptability curves will be generated to assess the probability of the TP being cost-effective at various willingness-to-pay thresholds.

ELIGIBILITY:
Inclusion criteria:

For participants in the intervention group (IG):

* 17 years old;
* diagnosed with type 1 diabetes, asthma and/or obesity;
* who had at least one pediatric outpatient visit, prior to inclusion, in one of both hospitals within the past 12 months;
* are Dutch speaking;
* planned to transfer to adult care within the next 12 months.

For participants in the control group (CG):

* age 17,5 and 18 years old, as the control period has a shorter duration (4 months vs. 12 months)
* diagnosed with type 1 diabetes, asthma and/or obesity;
* who had at least one pediatric outpatient visit, prior to inclusion, in one of both hospitals within the past 12 months;
* are Dutch speaking;
* planned to transfer to adult care within the next 12 months.

Exclusion criteria:

Applicable for both CG and IG:

- patients with severe mental, cognitive or neurological problems will be excluded

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Readiness to transition - TRAQ 6.0 | 12 months
  The TRAQ 6.0 (Transition Readiness Assessment Questionnaire version 6.0) is a tool designed to assess the readiness of youth with special healthcare needs to transition from pediatric to adult healthcare systems. It evaluates self-management and self-advocacy skills across key domains. The TRAQ 6.0 Dutch Version will be used. The TRAQ 6.0 has 20 items, with a theoretical range from 20 to 100. High TRAQ scores indicate a high level of transition readiness reflecting the individual demonstrates strong self-management and self-advocacy skills, such as managing medications, appointments, insurance, and understanding their own medical condition. Higher scores suggest the youth may be ready or nearly ready for transition to adult care. Low TRAQ scores indicate low transition readiness, indicating that the youth may lack knowledge or confidence in managing aspects of their healthcare, this reflects a need for additional support, education, or targeted transition planning.

SECONDARY OUTCOMES:
Generic Youth Patient Empowerment Scale (GYPES) | 12 months
  The Generic Youth Patient Empowerment Scale (GYPES) is a 15-item questionnaire designed to assess the level of empowerment in young patients with chronic conditions. Using a 5-point Likert scale, it yields a total score ranging from 15 to 75. Higher scores reflect greater empowerment, indicating that the young person feels more knowledgeable, confident, and involved in managing their healthcare, while lower scores suggest a need for additional support to strengthen self-management and engagement.
Morisky Medication Adherence Scale (MMAS) | 12 months
  The Morisky Medication Adherence Scale (MMAS) is a self-reported questionnaire designed to assess a patient's adherence to prescribed medication. It includes 8 items, with scores ranging from 0 to 8. Higher scores indicate better medication adherence, while lower scores suggest potential issues with taking medications as prescribed and may signal the need for interventions to improve adherence.
EQ-5D-5L | 12 months
  The EQ-5D-5L is a standardized questionnaire used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels of severity, and responses are combined into a single health profile that can be converted into an index score, typically ranging from less than 0 (representing health states worse than death) to 1 (representing full health). Higher scores reflect better perceived quality of life, while lower scores indicate greater health-related challenges.
Hospital Anxiety and Depression Scale (HADS) | 12 months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire used to assess levels of anxiety and depression in individuals with physical health problems. It consists of two subscales-anxiety and depression-each with 7 items, scored from 0 to 21. Higher scores indicate greater levels of anxiety or depression, with scores of 0-7 considered normal, 8-10 borderline, and 11-21 indicating clinically significant symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium